CLINICAL TRIAL: NCT03011268
Title: Continuing or Discontinuing Anti-tumor Necrosis Factor Treatment in Patients With Ulcerative Colitis in Clinical Remission: a Prospective Open Randomized Parallel-group Study
Brief Title: Anti-tumor Necrosis Factor in Patients With Ulcerative Colitis in Clinical Remission: to Continue or Not?
Acronym: BIOSTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Oslo University Hospital (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR2016-0.6; 2016-001409-18 (EudraCT Number)
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Colitis,Ulcerative
Keywords: Tumor Necrosis Factor-alpha/antagonists & inhibitors; Infliximab; Adalimumab; Golimumab; Recurrence
MeSH Terms: conditions — Colitis, Ulcerative; Recurrence | interventions — Infliximab; CT-P13; Adalimumab; golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti TNF discontinuation (Experimental): Discontinuation of anti-TNF treatment (Infliximab, Adalimumab, Golimumab)
  Interventions: Other: Discontinuation of anti-TNF treatment
- Anti TNF continuation (Active Comparator): Continuation of anti-TNF treatment (Infliximab, Adalimumab, Golimumab)
  Interventions: Other: Continuation of anti-TNF treatment

INTERVENTIONS:
Other: Discontinuation of anti-TNF treatment — Discontinuation of treatment with Infliximab, Adalimumab, and Golimumab in order to record time to relapse occurrences
  Other Names: Remicade, Remsima, Inflectra, Humira, Simponi
  Arms: Anti TNF discontinuation
Other: Continuation of anti-TNF treatment — Continuation of treatment with Infliximab, Adalimumab, and Golimumab for 2 years after randomization, then discontinue
  Other Names: Remicade, Remsima, Inflectra, Humira, Simponi
  Arms: Anti TNF continuation

SUMMARY:
The primary objective is to assess if discontinuation of anti- tumor necrosis factor alpha (TNF) treatment in ulcerative colitis patients in sustained clinical remission, with the option to restart treatment in the case of relapse, is non-inferior to continued anti-TNF treatment. Secondary objectives are to assess the efficacy and safety of restarting anti-TNF treatment after a relapse

DETAILED DESCRIPTION:
The BIOSTOP study is a prospective, open randomized, multicenter, parallel-group study to compare clinical outcome of discontinuing (interventional group) compared to continuing (control group) biologic treatment with anti-TNF in ulcerative colitis patients in clinical remission.

Adult male and female patients with an established diagnosis of ulcerative colitis treated for minimum one year with anti-TNF maintenance therapy and being in clinical remission during the last 3 months are potential study patients. Eligible patients who have given their informed written consent will be randomized 1:1 to either discontinue anti-TNF treatment or to continue anti-TNF treatment for another two years.

Patients in the control group who are still in clinical and endoscopic remission after two years on continued anti-TNF treatment, will then be switched to discontinue anti-TNF treatment.

End of study/follow-up is after 4 years. In order to identify the primary endpoint (occurrence of disease relapse), each study center will have a phone number for patients to call in case of symptoms suspect of increased disease activity. If a patient is experiencing a potential disease flare (6-point Mayo score > 1) and/or 2 consecutive calprotectin tests are positive (> 200 mg/kg), an unscheduled visit including recto sigmoidoscopy will be performed without delay to document disease status.

150 participants enrolled, September 2020 Covid 19 - randomization period extended until 31.12.2020

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of ulcerative colitis
* treated for minimum 1 year with first-line anti-tumor necrosis factor (TNF) treatment
* in sustained clinical remission during the last 3 months
* capable of understanding and signing an informed consent form

Exclusion Criteria:

* Discontinuation of systemic 5-Aminosalicylic acid (ASA) or immunomodulatory therapy or other medication that could affect disease activity during the last 3 months prior to randomization
* Any treatment of systemic corticosteroids due to disease exacerbation during the last 3 months (i.e. patients being in steroid free clinical remission)
* Patients on anti-TNF monotherapy with intolerance to both 5-ASA and immunomodulatory therapy
* Change in the anti-TNF treatment during the last 3 months due to disease related factors, not including dose/frequency adjustments due to drug concentration measurements
* Use of any second-line anti-TNF medication irrespective of reason for stopping first-line anti-TNF
* Previous failed attempts of anti-TNF discontinuation of more than 4 months' duration, with the exception of discontinuation due to pregnancy
* Detection of anti-TNF antibodies in moderate-high titers prior to randomization
* Psychiatric or mental disorders
* Alcohol abuse or other substance abuse
* language barriers or other factors which makes adherence to the study protocol impossible
* Participation in any other studies
* pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in sustained clinical remission | 2 years
  Remission confirmed endoscopically by mucosal healing defined as Mayo Endoscopic Subscore (MES) score 0 or 1 after 2 years of randomized treatment

SECONDARY OUTCOMES:
Proportion of patients in sustained clinical remission | 4 years
  Remission confirmed endoscopically by mucosal healing defined as Mayo Endoscopic Subscore (MES) score 0 or 1 after 4 years of randomized treatment
Time from randomization to relapse | 2 years
  Relapse time
Time from randomization to relapse | 4 years
  Relapse time
Proportion of patients who are no longer in remission, but who do not need to restart anti-tumor necrosis factor (TNF) therapy | 2 years
  Remission, but no need to restart anti-tnf therapy
Proportion of patients who are no longer in remission, but who do not need to restart anti-tumor necrosis factor (TNF) therapy | 4 years
  Remission, but no need to restart anti-tnf therapy
Proportion of relapse patients achieving remission after anti-TNF restart | 2 years
  Remission after relapse
Proportion of relapse patients achieving remission after anti-TNF restart | 4 years
  Remission after relapse
Adverse events and serious adverse events frequency and severity | 2 years
  Adverse events
Adverse events and serious adverse events frequency and severity | 4 years
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dag Arne L Hoff, md, phd, Study Director — Helse Møre og Romsdal Hospital Trust
Locations (19):
- Norway (19):
  - Helse Møre og Romsdal, Ålesund Sjukehus, Ålesund
  - Haraldsplass Diakonale sykehus, Bergen
  - Haukeland Universitetssykehus Helse Bergen HF, Bergen
  - Sykehuset Østfold HF Kalnes, Fredrikstad
  - Helse Førde, Førde Sentralsjukehus, Førde
  - Sykehuset Innlandet, Hamar Sykehus, Hamar
  - Universitetssykehuset i Nord-Norge, Harstad, Harstad
  - Sørlandet Sykehus HF, Kristiansand, Kristiansand
  - Helse Møre og Romsdal, Kristiansund Sjukehus, Kristiansund
  - Helse Nord Trøndelag, Levanger Sykehus, Levanger
  - Akershus Universitetssykehus, Lørenskog, Lørenskog
  - Oslo Universitetssykehus, Rikshospitalet, Oslo
  - Oslo Universitetssykehus, Ullevål, Oslo
  - Vestre Viken HF, Bærum Sykehus, Sandvika
  - Sykehuset Telemark, Skien, Skien
  - Stavanger Universitetssykehus, Stavanger
  - Sykehuset Vestfold, Tønsberg, Tønsberg
  - Helse Møre og Romsdal, Volda Sjukehus, Volda
  - Helse Bergen HF Voss Sjukehus, Voss

IPD SHARING:
Plan to Share IPD: No
At this time there is no such plan for IPD sharing. It might be an issue regarding material stored in the study Biobank - that will be elucidated at a later stage.